CLINICAL TRIAL: NCT03445039
Title: Clinical Evaluation of Modified Transalveolar Sinus Floor Elevation and Osteotome Sinus Floor Elevation in Posterior Maxillae
Brief Title: Clinical Evaluation of Two Types of Transalveolar Sinus Floor Elevation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xu Zhao, clinician, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: modified maxillary sinus lift
Record Dates: First submitted 2018-01-25; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Dental Implant; Sinus Floor Augmentation
Keywords: Dental implants, Trans-alveolar sinus floor elevation, Bone grafting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All of the patients will be divided into four groups by using randomization tables. The assignment will be concealed from the clinical operators until the beginning of implant surgery. The outcome examiners will be kept blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TSFE using osteotomes with bone grafting (Experimental): The patients in this group will receive transalveolar sinus floor elevation with osteotomes and mallet. The bone substitute is placed in this group.The interventions in the arm are bone grafting and the TSFE will be performed by osteotomes.
  Interventions: Device: traditional TSFE; Procedure: bone grafting materials
- TSFE using osteotomes without bone grafting (Experimental): The patients in this group will receive transalveolar sinus floor elevation with osteotomes and mallet. The bone substitute will not be placed in this group.The intervention in the arm is the TSFE will be performed by osteotomes.
  Interventions: Device: traditional TSFE; Procedure: without bone grafting materials
- modified TSFE with bone grafting (Experimental): The patients in this group will receive modified transalveolar sinus floor elevation with the Dask drills. The cortical plate of the sinus floor is grinded or removed by the dome like drills. And the membrane is elevated by the surgical instruments. The bone substitute is placed before the implant placement.Interventions in the arm are bone grafting and the TSFE will be performed by dask drills.
  Interventions: Procedure: bone grafting materials; Device: TSFE by DASK drills
- modified TSFE without bone grafting (Experimental): The patients in this group will receive modified transalveolar sinus floor elevation with the Dask drills. The cortical plate of the sinus floor is grinded or removed by the dome like drills. And the membrane is elevated by the surgical instruments. The bone substitute will not be placed in this group.The intervention in the arm is the TSFE will be performed by dask drills.
  Interventions: Device: TSFE by DASK drills; Procedure: without bone grafting materials

INTERVENTIONS:
Device: traditional TSFE — The TSFE procedure is performed by osteotomes (Straumann AG, Basel, Switzland) and mallet as the traditional ways.
  Arms: TSFE using osteotomes with bone grafting; TSFE using osteotomes without bone grafting
Procedure: bone grafting materials — The bone substitute is placed into the siuns under the membrane before the implant placement
  Arms: TSFE using osteotomes with bone grafting; modified TSFE with bone grafting
Device: TSFE by DASK drills — The TSFE procedure is performed by DASK(Dentium Advanced Surgical Kits) drills (Dentium, Korea), the residual cortical plate of the sinus floor is grinded by the drills.
  Arms: modified TSFE with bone grafting; modified TSFE without bone grafting
Procedure: without bone grafting materials — The bone substitute will not be placed into the sinus before the implant placement.
  Arms: TSFE using osteotomes without bone grafting; modified TSFE without bone grafting

SUMMARY:
Background: Implant placement in the posterior maxilla is always troubled by the insufficient bone volume. Trans-alveolar sinus floor elevation (TSFE) has been proven a predictable surgical procedure to increase the bone height in the posterior maxilla. However, questions as the necessity of the bone grafting is necessary during the sinus lift and could the TSFE be performed when the residual bone height is below 5mm are still being debated. Besides, high-quality evidence on comparing the clinical outcome of transalveolar sinus floor elevation with osteotome and modified sinus floor elevation with crestal non-cutting drills is limited.

Methods/Design: 120 adult patients who fit the inclusion criterions are being recruited from the first clinical division, School and Hospital of Peking University (Beijing, China). All the patients are assigned into four groups according a table of random numbers. Participants receive 1) TSFE using osteotomes with bone grafting; 2) TSFE using osteotomes without bone grafting; 3) modified TSFE with bone grafting; and 4) modified TSFE without bone grafting. The clinical operators will be concealed with the assignment until the beginning of surgical procedures. In a one year follow up period, implant survival rates, complications, implant stability, bone remodeling around the implant and patient-reported outcome (visual analogue scale for intraoperative discomfort and postoperative pain) are observed and documented. The implant stability is gauged by the resonance frequency analysis for 7 times (2, 4,8,12,16,26,52 weeks). And the bone remodeling is observed and compared by CT scan.

Discussion: The result of the trial will support a better decision making in atrophy posterior maxilla when implant placement is needed. If favorable, the use of the modified TSFE would achieve as ideal outcome as the traditional TSFE but with less trauma and postoperative discomforts. Besides, whether the bone graft procedure is necessary for the TSFE will also be discussed.

ELIGIBILITY:
Inclusion Criteria:

* patients who is more than 18 years old;
* patients have lost a single tooth or several teeth in the posterior area of the maxilla, the tooth has/have been extracted for more than three months;
* The residual bone height was between 3mm to 6mm;
* The width of the alveolar ridge could contain the implant with standard diameter;
* The general and local status of patient are suitable for implant placement and sinus floor elevation;
* The patient who is willing to sign the informed consent and to follow the experimental follow-up rules.

Exclusion Criteria:

* Uncontrolled systemic diseases as diabetes, hypertension and so on;
* Uncontrolled local diseases as periodontal disease or muco- cutaneous disease;
* Heavy smoker (more than 10 cigarettes /day)
* Patients who is suffering rhinitis, sinusitis; or rather large cyst is found in the maxillary sinus
* The bone density of the maxillary posterior region is too poor to maintain the initial stability of the implant
* The target of the implant site once received implant therapy or bone grafting
* Patient with psychogenia or incapable to understand and obey the doctors' instruction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-02 (Actual); Primary Completion 2019-12-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
implant survival rate | the implant status will be inspected and calculated at 1 year revisit
  whether the implant has osseointegrated and functional
implant stability | 2 weeks after implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 4 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 8 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 12 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 16 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 26 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
implant stability | 52 weeks after the implant placement
  the implant stability is gauged by the RFA( resonance frequency analysis)
marginal bone remodeling around the implant | 26 weeks after the implant placement
  use CBCT to access the marginal bone changes between the 26 weeks after the implant placement and baseline (the day the implant is placed).
marginal bone remodeling around the implant | 52 weeks after the implant placement
  use CBCT to access the marginal bone changes between the 52 weeks after the implant placement and baseline (the day the implant is placed).
post operative pain accessed by the patient | 1 day after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 2 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 3 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 4 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 5 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 6 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 7 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative pain accessed by the patient | 14 days after the surgery
  The post operative pain is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No pain" and "worst imaginable pain". The patient will mark on the line to represent their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 1 day after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 2 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 3 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 4 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 5 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 6 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 7 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.
post operative swelling accessed by the patient | 14 days after the surgery
  The post operative swelling is access by the patient via visual analog scales. The VAS questionnaire consists a 100mm long and two anchors, one at each end. The anchors are verbal "No swelling" and "worst imaginable swelling". The patient will mark on the line to represent their swelling intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no swelling" anchor and the patient's mark, providing a range of scores from 0-100.

SECONDARY OUTCOMES:
sulcus bleeding around the implant | 26 weeks after the implant placement
  the sulcus bleeding index is used to measure whether there is bleeding when the dental prob is inserte the sulcus around the implant site
dental plaque around the implant | 26 weeks after the implant placement
  measure whether there is dental plaque around the implant
other complications | through study completion, up to 1 year
  including post-operative infection, bleeding in the nostril,hematoma, stuffy nose and benign paroxysmal positional vertigo
sulcus bleeding around the implant | 52 weeks after the implant placement
  the sulcus bleeding index is used to measure whether there is bleeding when the dental prob is inserte the sulcus around the implant site
dental plaque around the implant | 52 weeks after the implant placement
  measure whether there is dental plaque around the implant

CONTACTS AND LOCATIONS:
Overall Officials: Feng Liu, Dr, Study Director — Peking University hospital of stomatology, the first clinical division
Locations (1):
- Peking University, Hospital of stomatology, the first clinical division, Beijing, China

REFERENCES:
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Summers RB. The osteotome technique: Part 3--Less invasive methods of elevating the sinus floor. Compendium. 1994 Jun;15(6):698, 700, 702-4 passim; quiz 710. PMID 7994726
- [Background] Lozada JL, Goodacre C, Al-Ardah AJ, Garbacea A. Lateral and crestal bone planing antrostomy: a simplified surgical procedure to reduce the incidence of membrane perforation during maxillary sinus augmentation procedures. J Prosthet Dent. 2011 Mar;105(3):147-53. doi: 10.1016/S0022-3913(11)60020-6. PMID 21356405
- [Background] French D, Nadji N, Shariati B, Hatzimanolakis P, Larjava H. Survival and Success Rates of Dental Implants Placed Using Osteotome Sinus Floor Elevation Without Added Bone Grafting: A Retrospective Study with a Follow-up of up to 10 Years. Int J Periodontics Restorative Dent. 2016;36 Suppl:s89-97. doi: 10.11607/prd.2191. PMID 27031637
- [Result] Tan WC, Lang NP, Zwahlen M, Pjetursson BE. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. Part II: transalveolar technique. J Clin Periodontol. 2008 Sep;35(8 Suppl):241-54. doi: 10.1111/j.1600-051X.2008.01273.x. PMID 18724853
- [Result] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Result] Markovic A, Misic T, Calvo-Guirado JL, Delgado-Ruiz RA, Janjic B, Abboud M. Two-Center Prospective, Randomized, Clinical, and Radiographic Study Comparing Osteotome Sinus Floor Elevation with or without Bone Graft and Simultaneous Implant Placement. Clin Implant Dent Relat Res. 2016 Oct;18(5):873-882. doi: 10.1111/cid.12373. Epub 2015 Aug 28. PMID 26315564
- [Result] Caban J, Fermergard R, Abtahi J. Long-term evaluation of osteotome sinus floor elevation and simultaneous placement of implants without bone grafts: 10-Year radiographic and clinical follow-up. Clin Implant Dent Relat Res. 2017 Dec;19(6):1023-1033. doi: 10.1111/cid.12530. Epub 2017 Aug 29. PMID 28853214
- [Derived] Zhao X, Gao W, Liu F. Clinical evaluation of modified transalveolar sinus floor elevation and osteotome sinus floor elevation in posterior maxillae: study protocol for a randomized controlled trial. Trials. 2018 Sep 14;19(1):489. doi: 10.1186/s13063-018-2879-x. PMID 30217227